CLINICAL TRIAL: NCT01687829
Title: Macular Hole Surgery With and Without Internal Limiting Membrane Peeling：A Systematic Review and Meta-analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yifan Feng (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Yifan Feng, Eye Hospital, Wenzhou Medical College, China, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: F20120913
Record Dates: First submitted 2012-09-13; First posted 2012-09-19 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Macular Holes
Keywords: Macular Holes; Internal limiting membrane; peeling; Surgery
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- ILM-on group: patients were scheduled to undergo macular hole surgery without internal limiting membrane (ILM) peeling
- ILM-off group: patients were scheduled to undergo macular hole surgery with internal limiting membrane (ILM) peeling

SUMMARY:
Since Kelly and Wendel first reported successful closure of idiopathic macular holes (MH) by vitrectomy in 1991, many surgical modifications have been made to improve the anatomical and visual outcomes of this surgery. Recently, internal limiting membrane (ILM) peeling has become used widely as an adjunctive procedure during MH surgery because the removal of ILM is thought to reduce the tangential traction on the macula, a major factor in the pathogenesis of idiopathic macular holes. However, the role of ILM peeling in macular hole surgery is not yet well defined. To the best of our knowledge, there is no meta-analysis on comparison of the efficacy of ILM peeling and suture for MH surgery. This study reviewed the published literature comparing surgical results with and without ILM peeling and and performed a meta-analysis to determine whether there is any benefit or detriment anatomically and/or visually.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are those with idiopathic FTMH in stages 2-3, of less or equal than 18 months duration (based on symptoms reported by the patient) and with a visual acuity equal to or worse than 20/40 in the study eye.

Exclusion Criteria:

* Patients with idiopathic FTMH stages 2-3 but longer than 18 months duration or with other causes of decreased vision (e.g. corneal scarring, age-related macular degeneration, diabetic retinopathy, glaucoma if central and/or paracentral absolute visual field defects are present) and
* Those with FTMH related to high myopia (> 6 dioptres) or trauma will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients were scheduled to undergo macular hole surgery and randomized to with and without internal limiting membrane (ILM) peeling
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Anatomic Success rate | 12 months
  Anatomic success defined as a closed hole without a visible edge or a flat hole without a rim of subretinal fluid.
Functional Success Rate | 12 month
  Functional Success defined as an improvement of 2 or more Snellen BCVA.

SECONDARY OUTCOMES:
Best-corrected visual acuity | 12 month
  All Snellen BCVA were converted to logarithm of the minimum angle of resolution (logMAR) BCVA
Complications | 12 months
  Such as elevated intraocular pressure,retinal tear,rhegmatogenous retinal detachment

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Feng, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China